CLINICAL TRIAL: NCT00180492
Title: Carotid RX ACCULINK(TM)/ACCUNET(TM) Post-Approval Trial to Uncover Unanticipated or Rare Events - CAPTURE
Brief Title: Post-Approval Study of the Guidant Carotid Stent Systems and Embolic Protection Systems: CAPTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Guidant Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 04-715
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Atherosclerotic Disease, Carotid
Keywords: Atherosclerotic disease
MeSH Terms: conditions — Carotid Artery Diseases

INTERVENTIONS:
Device: RX ACCULINK(TM) Carotid Stent System and RX ACCUNET(TM) Embolic Protection System

SUMMARY:
This purpose of this study is to collect data on the FDA-approved ACCULINK(TM) Carotid Stent System and FDA 510(k)-cleared ACCUNET(TM) Embolic Protection System for the treatment of patients with atherosclerotic disease, when used by physicians under commercial use conditions.

DETAILED DESCRIPTION:
CAPTURE is a post-approval study to collect information on the safety and effectiveness of the ACCULINK and ACCUNET since the approval/clearance of these devices by the FDA. The ACCULINK stent is an elastic-like metal tube that is used to hold open a narrow part of a blood vessel. The ACCUNET is a wire mesh basket that is placed in the vessel to catch material (blood clots, fatty material) that could break off from the narrowed area of the blood vessel and block blood flow downstream during the stent procedure.

Another goal of the CAPTURE study is to confirm that the ACCULINK and ACCUNET can be used safely by physicians with varying levels of experience in stenting procedures.

The basis for FDA's approval/clearance of the ACCULINK and ACCUNET was the ARCHeR trials (ACCULINK/ACCUNET for Revascularization of Carotids in High-Risk Patients). The ARCHeR trials were conducted to collect data on the safety and effectiveness of the ACCULINK and ACCUNET when used in the treatment of carotid artery disease in patients at high risk for surgical treatment (carotid endarterectomy) because of medical or surgical comorbidities. The ARCHeR trials showed that the ACCULINK, used with or without the ACCUNET, is a safe and effective treatment option based on the rate of death, stroke, and myocardial infarction at 30 days, and stroke at one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient's physician used an ACCULINK and/or ACCUNET

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Death, stroke, and myocardial infarction at 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Walker, PhD, Study Chair — Abbott Medical Devices
Locations (1):
- Guidant Corporation, Santa Clara, California, United States